CLINICAL TRIAL: NCT01806064
Title: A Randomized Phase 2 Trial of Axitinib and TRC105 Versus Axitinib Alone (Including a lead-in Phase 1B Dose Escalation Portion) in Patients With Advanced or Metastatic Renal Cell Carcinoma
Brief Title: Randomized Phase 2 Trial of Axitinib and TRC105 Versus Axitinib Alone in Patients Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study did not meet endpoint.
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105RC101
Record Dates: First submitted 2013-02-26; First posted 2013-03-07 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Renal Cell Carcinoma
Keywords: TRC105; CD105; RCC; Renal Cell Carcinoma; Axitinib; INLYTA; Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — carotuximab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRC105 and Axitinib (Experimental): Patients randomized to receive TRC105 at 3 mg/kg on day 1, 7 mg/kg on day 4, and 10 mg/kg on day 8 and weekly thereafter in combination with axitinib 5 mg twice daily
  Interventions: Drug: TRC105 and Axitinib
- Axitinib (Active Comparator): Patients randomized to receive axitinib 5 mg twice daily
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: TRC105 and Axitinib
  Other Names: Chimeric Antibody (TRC105) to CD105; Inlyta
  Arms: TRC105 and Axitinib
Drug: Axitinib
  Other Names: Inlyta
  Arms: Axitinib

SUMMARY:
Phase 1b: To evaluate safety and tolerability and determine a recommended phase 2 dose for TRC105 when added to standard dose axitinib in patients with advanced renal cell carcinoma.

Phase 2: To estimate the PFS of patients with advanced or metastatic RCC by RECIST 1.1 criteria in patients treated with axitinib and TRC105 compared to those treated with axitinib alone, following failure of one prior VEGF TKI

DETAILED DESCRIPTION:
Axitinib is an oral inhibitor of multiple receptor tyrosine kinases including vascular endothelial growth factor receptor VEGFR-1, VEGFR-2, and VEGFR-3 at therapeutic plasma concentrations. These receptors are implicated in pathologic angiogenesis, tumor growth, and cancer progression. Axitinib is approved for the treatment of advanced renal cell carcinoma, following progression on one prior systemic therapy. TRC105 is an antibody to CD105, an important angiogenic target on vascular endothelial cells that is distinct from VEGFR. TRC105 inhibits angiogenesis, tumor growth and metastases in preclinical models and complements the activity of bevacizumab and multi-kinase inhibitors that target VEGFR. In a phase 1 study of advanced solid tumors,TRC105 therapy caused a global reduction in angiogenic biomarkers and reduced tumor burden at doses that were well-tolerated. By targeting a non-VEGF pathway that is upregulated following VEGF inhibition, TRC105 has the potential to complement VEGF inhibitors and could represent a major advance in cancer therapy. TRC105 potentiates bevacizumab and VEGFR tyrosine kinases (VEGFR TKI) in preclinical models. In a phase 1b study, the combination of TRC105 and bevacizumab produced radiographic reductions in tumor volume in bevacizumab refractory patients. Together, the use of TRC105 with axitinib may result in more effective angiogenesis inhibition and improved clinical efficacy over that seen with axitinib alone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced or metastatic renal cell carcinoma with a clear cell component that has progressed by investigator assessment following treatment with one and only one multi-targeted tyrosine kinase inhibitor (TKI) other than axitinib that targets the VEGF receptor (VEGFR) (e.g., sunitinib, pazopanib, sorafenib, tivozanib, cabozantinib). One prior immunotherapy (interleukin-2 or interferon-alpha or immune checkpoint inhibitor or tumor vaccine) and one prior mTOR inhibitor treatment are allowed.
2. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission per investigators' clinical judgment.
3. Measurable disease by RECIST 1.1 criteria
4. Age of 18 years or older
5. ECOG performance status ≤ 1
6. Resolution of all acute adverse events resulting from prior cancer therapies to NCI CTCAE grade ≤ 1 or baseline (except alopecia)
7. Adequate organ function as defined by the following criteria:
8. Willingness and ability to consent for self to participate in study
9. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

1. Prior treatment with TRC105 or axitinib or any agent targeting the endoglin pathway (including a fusion protein that binds bone morphogenic protein)
2. Grade 3 or 4 toxicity related to prior VEGFR TKI that did not resolve to grade 1
3. Current treatment on another therapeutic clinical trial
4. Receipt of a small molecule anticancer agent, including an investigational anticancer small molecule, within 14 days of starting study treatment or receipt of a biologic anticancer agent (e.g., antibody) within 28 days of starting study treatment.
5. Prior radiation therapy within 28 days of starting the study treatment, except radiation therapy for bone metastases or radiosurgery is permitted up to 14 days of starting treatment
6. No major surgical procedure or significant traumatic injury within 6 weeks prior to study registration, and must have fully recovered from any such procedure; date of surgery (if applicable). Note: the following are not considered to be major procedures and are permitted up to 7 days before therapy initiation: Thoracentesis, paracentesis, port placement, laparoscopy, thorascopy, tube thoracostomy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, incisional biopsies, imaging-guided biopsy for diagnostic purposes, and routine dental procedures
7. Uncontrolled chronic hypertension defined as systolic > 150 or diastolic > 90 despite optimal therapy (initiation or adjustment of BP medication prior to study entry is allowed provided that the average of 3 BP readings at a visit prior to enrollment is < 150/90 mm Hg)
8. History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease. Patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered for at least 28 days.
9. Angina, MI, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, PTCA or CABG within the past 6 months. Deep venous thrombosis within 6 months unless the patient is anticoagulated without the use of warfarin for at least 2 weeks. In this situation, low molecular weight heparin is preferred.
10. Active bleeding or pathologic condition that carries a high risk of bleeding (e.g. hereditary hemorrhagic telangiectasia).
11. Thrombolytic use (except to maintain i.v. catheters) within 10 days prior to first day of study therapy
12. Known active viral or nonviral hepatitis or cirrhosis
13. History of hemorrhage or hemoptysis (> ½ teaspoon bright red blood) within 3 months of starting study treatment
14. History of peptic ulcer disease within 3 months of treatment, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 28 days of starting study treatment
15. History of gastrointestinal perforation or fistula in the past 6 months, or while previously on antiangiogenic therapy, unless underlying risk has been resolved (e.g., through surgical resection or repair)
16. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
17. Requirement for concomitant medications that strongly induce or inhibit CYP3A4/5
18. Pregnancy or breastfeeding. Female patients must be surgically sterile (i.e.: hysterectomy) or be postmenopausal, or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. All female patients of reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to first dose. Male patients must be surgically sterile or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. The definition of effective contraception will be based on the judgment of the Principal Investigator or a designated associate.
19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD PhD, Study Director — ctheuer@traconpharma.com
Locations (39):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - University of California, Irvine, Irvine, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Illinois CancerCare, Peoria, Illinois
  - Indiana Univeristy, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Atlantic Health System, Morristown, New Jersey
  - Gabrail Cancer Center Research, Canton, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - University of Utah, Salt Lake City, Utah
- Czechia (5):
  - Masaryk Institute, Brno
  - St. Anne's, Brno
  - University Hospital Brno, Brno
  - Na Bulovce Hospital, Prague
  - Thomayer Hospital, Prague
- Hungary (5):
  - Integrated Szent Istvan and Szent Laszlo Hospital, Budapest
  - National Institute of Oncology, Budapest
  - University of Debrecen Medical Center Institute of Oncology, Debrecen
  - Kaposi Mor Teaching Hospital, Kaposvár
  - Medical Center of the University of Pecs, Pécs
- Sussex Cancer Center, Royal Sussex County Hospital, Brighton, East Sussex, United Kingdom

REFERENCES:
- [Derived] Choueiri TK, Michaelson MD, Posadas EM, Sonpavde GP, McDermott DF, Nixon AB, Liu Y, Yuan Z, Seon BK, Walsh M, Jivani MA, Adams BJ, Theuer CP. An Open Label Phase Ib Dose Escalation Study of TRC105 (Anti-Endoglin Antibody) with Axitinib in Patients with Metastatic Renal Cell Carcinoma. Oncologist. 2019 Feb;24(2):202-210. doi: 10.1634/theoncologist.2018-0299. Epub 2018 Sep 6. PMID 30190302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 patients enrolled in phase 1b portion. 150 patients randomized in the phase 2 portion.
Groups:
- P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID: Phase 1b Dose Level 1: 8 mg/kg TRC105 weekly in combination with 5 mg Axitinib twice daily
- P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID: Phase 1b Dose Level 2: 10 mg/kg TRC105 weekly in combination with 5 mg Axitinib twice daily
- P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID: Phase 1b Dose Level 3: 10 mg/kg TRC105 weekly during cycle 1 then 15 mg/kg TRC105 every two weeks beginning in cycle 2 in combination with 5 mg Axitinib twice daily
- P2 Arm A: 5 mg Axitinib BID: Phase 2 Arm A: 5 mg Axitinib twice daily
- P2 Arm B: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID: Phase 2 Arm B: 10 mg/kg TRC105 weekly + 5 mg Axitinib twice daily
Period: Overall Study
Arm/Group | P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID | P2 Arm A: 5 mg Axitinib BID | P2 Arm B: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID
Started | 3 | 15 | 5 | 75 | 75
Completed | 3 | 15 | 5 | 74 | 73
Not Completed | 0 | 0 | 0 | 1 | 2
Not completed — Randomized Not Enrolled | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All patients who received at least a portion of a dose of TRC105 or axitinib
Groups:
- Total: Total of all reporting groups
Arm/Group | P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID | P2 Arm A: 5 mg Axitinib BID | P2 Arm B: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID | Total
Number analyzed (Participants) | 3 | 15 | 5 | 75 | 75 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 13 | 2 | 35 | 43 | 93
  >=65 years | 3 | 2 | 3 | 40 | 32 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 18 | 26 | 48
  Male | 3 | 13 | 3 | 57 | 49 | 125
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3 | 12 | 5 | 70 | 71 | 161
  Hispanic or Latino | 0 | 3 | 0 | 5 | 1 | 9
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 0 | 0 | 0 | 11 | 10 | 21
  United States | 3 | 15 | 5 | 56 | 59 | 138
  Czechia | 0 | 0 | 0 | 8 | 5 | 13
  United Kingdom | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Patients With DLT
Description: Phase 1b: For dose limiting toxicity (DLT) evaluation, severity (grade) was classified according to common terminology criteria for adverse events version 4.0 (CTCAE v4.0).
Time Frame: 12 Months
Population: Patients who discontinued the study prior to completing the DLT evaluation period were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID
Number analyzed (Participants) | 3 | 15 | 5
Participants | 0 | 0 | 0

2. Primary Outcome: Phase 2: Progression Free Survival (PFS) of Patients With RCC
Description: Median progression free survival (PFS) of patients with advanced or metastatic RCC by RECIST 1.1. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 15 Months
Population: 95% confidence interval was applied. "NA" is listed for the confidence interval if there were not enough events to estimate a standard error. For Phase 2 all randomized patients were included in the efficacy population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | P2 Arm A: 5 mg Axitinib BID | P2 Arm B: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID
Number analyzed (Participants) | 75 | 75
Months | 11.4 [5.8 to NA] — Confidence interval was not estimable if there were not enough events to estimate a standard error. | 6.7 [5.6 to 13.1]

3. Secondary Outcome: Phase 1b & 2: Response Rate of Patients With RCC
Description: Number of patients with partial response (PR) or complete response (CR) by RECIST 1.1 criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 15 Months
Population: For Phase 1b patients with screening and at least one on study scan were included in the efficacy population. For Phase 2 all randomized patients were included in the efficacy population. Patients without a baseline scan and at least 1 on study scan were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P2 Arm A: 5 mg Axitinib BID | P2 Arm B: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID
Number analyzed (Participants) | 3 | 75 | 75 | 14 | 5
Participants | 0 | 22 | 23 | 5 | 0

4. Secondary Outcome: Phase 2: Overall Response Rate of Patients With RCC by Choi
Description: Overall response (OR) rate is the number of patients with partial response (PR) or complete response (CR) by Choi Criteria. Per Choi criteria for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), A decrease in size ≥ 10% or a decrease in tumor attenuation (Houndsfield units) ≥ 15% on CT and no new lesions; Overall Response (OR) = CR + PR.
Time Frame: 15 Months
Population: For Phase 2 all randomized patients were included in the efficacy population. Patients without a baseline scan and at least 1 on study scan were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | P2 Arm A: 5 mg Axitinib BID | P2 Arm B: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID
Number analyzed (Participants) | 75 | 75
Participants | 50 | 50

5. Secondary Outcome: Phase 1b & 2: Trough Concentrations of TRC105 by Dose Level in Phase 1b
Description: Trough Serum TRC105 concentrations at steady state (cycle 2 day 15) were measured using validated ELISA methods.
Time Frame: 2.5 months (cycle 2 day 15)
Population: In 1b patients with a predose sample collected at cycle 2 day 15 were averaged. Patients who missed a dose of TRC105 prior to cycle 2 day 15 were excluded from the analysis. Additional Phase 1b PK analysis beyond steady state concentration at cycle 2 day 15 were not performed. Samples collected in the phase 2 portion of the study were not analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID
Number analyzed (Participants) | 3 | 13 | 5
ng/mL | 27650 (39103) | 140022 (45403.01) | 54375 (23546.5)

6. Secondary Outcome: Phase 1b & 2: Number of Patients With Development of Immunogenicity Antibodies.
Description: Anti-product antibody concentration were measured using validated ELISA methods.
Time Frame: 12 months
Population: Patients must have had a baseline and on study assessment of immunogenicity and their baseline must have been negative.
  Samples collected in the phase 2 portion of the study were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID
Number analyzed (Participants) | 3 | 5 | 5
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years, 6 months
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Only patients who received at least a portion of a dose of TRC105 and/or Axitinib have been included in the analysis population.
Arm/Group | P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID | P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID | P2 Arm A: 5 mg Axitinib BID | P2 Arm B: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/15 | 0/5 | 3/74 | 6/73
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/15 | 3/5 | 27/74 | 28/73
Other Adverse Events (participants affected / at risk) | 3/3 | 15/15 | 5/5 | 71/74 | 72/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID (N=3) | P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID (N=15) | P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID (N=5) | P2 Arm A: 5 mg Axitinib BID (N=74) | P2 Arm B: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID (N=73)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2 (3) | 0 (0)
Acute Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (8)
Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Biliary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal Vein Occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 0 | 1 | 0 | 0 (0) | 4 (4)
Clostridium Difficile Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 (0) | 0 (0)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 (0) | 3 (3)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Enterococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0)
Colonic Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ Failure (General disorders) | 0 | 1 | 0 | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumothroax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior Reversible Encephalopothy Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | P1b: 8 mg/kg TRC105 Wkly + 5 mg Axitinib BID (N=3) | P1b: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID (N=15) | P1b: 10 mg/kg Wkly/15 mg/kg q2wks TRC105 + 5 mg Axitinib BID (N=5) | P2 Arm A: 5 mg Axitinib BID (N=74) | P2 Arm B: 10 mg/kg TRC105 Wkly + 5 mg Axitinib BID (N=73)
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 3 | 0 | 3 | 1
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 5 | 1 | 2 | 10
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 11
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abnormal Dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 0 | 0 | 0 | 2
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 1 | 2
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 0 | 4 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 1 | 12 | 16
Anal Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Anorectal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 5 | 2
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 10 | 8
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 3 | 0 | 7 | 5
Asthenia (General disorders) | 3 | 2 | 0 | 9 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 17 | 7
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 3
Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bladder Spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 2 | 7
Blood Amylase Increased (Investigations) | 1 | 1 | 0 | 7 | 2
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 9 | 5
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 2 | 1
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 0 | 4 | 5
Blood Urea Increased (Investigations) | 0 | 0 | 0 | 2 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3
Brachycardia (Cardiac disorders) | 0 | 1 | 0 | 3 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bundle Branch Block Right (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Burning Sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Candidiasis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Cardiac Disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac Murmur (Investigations) | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 2 | 0
Catheter Site Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Catheter Site Swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerumen Impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chest Discomfort (General disorders) | 0 | 1 | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 2 | 0 | 4 | 1
Chills (General disorders) | 3 | 1 | 1 | 7 | 11
Choking Sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Colostomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 1 | 0 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 5 | 2 | 13 | 21
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary Artery Thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 15 | 14
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 3
Dacryocanaliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 5 | 3 | 26 | 21
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0 | 7 | 11
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 2 | 4
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 11 | 4 | 46 | 42
Diarrhoea Infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diastolic Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Disturbance In Attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 1 | 9 | 10
Dizziness Postural (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Drug Intolerance (General disorders) | 0 | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 7 | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 4
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 9 | 10
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dyskinesia Oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 10 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 3 | 27 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 10 | 12
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3 | 3
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ear Discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 3
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 0 | 0 | 3
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Epidermal Growth Factor Receptor Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 13 | 5 | 5 | 47
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 6
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye Pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Facial Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Faecal Incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Faeces Discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Faeces Pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 4
Fatigue (General disorders) | 3 | 9 | 4 | 40 | 42
Feeling Cold (General disorders) | 0 | 1 | 0 | 0 | 1
Feeling Hot (General disorders) | 0 | 0 | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 5
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 7
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 7
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Food Intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fungal Skin Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Gallbladder Pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 3
Genital Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 1
Gingival Bleeding (Gastrointestinal disorders) | 2 | 7 | 5 | 3 | 25
Gingival Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Glucose Urine Present (Investigations) | 0 | 0 | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 8
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 8
Haemoglobin Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 4
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 10 | 2 | 12 | 47
Hearing Impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hyperaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 5 | 2
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 6 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 4 | 4 | 33 | 26
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 5 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 6 | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 2 | 7
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 20 | 17
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 3
Incision Site Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 3 | 2
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 19
Infusion Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Infusion Site Extravasation (General disorders) | 0 | 0 | 0 | 0 | 1
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Inguinal Mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Injection Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Injection Site Haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1
Injection Site Mass (General disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 1 | 6 | 5
International Normalised Ratio Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Iron Binding Capacity Total Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 2
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 2 | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Lipase Increased (Investigations) | 1 | 1 | 0 | 5 | 2
Livedo Reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Liver Disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Liver Function Test Increased (Investigations) | 0 | 1 | 0 | 1 | 0
Local Swelling (General disorders) | 0 | 0 | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lymph Gland Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1 | 4 | 3
Medical Device Site Bruise (General disorders) | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Mental Impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Metabolic Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 5
Mitral Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 7 | 0 | 6 | 10
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3 | 2
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4 | 4
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 6 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 5 | 7
Mycobacterium Tuberculosis Complex Test Positive (Investigations) | 0 | 0 | 0 | 0 | 1
Nail Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Nail Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 6
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Nasal Septum Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal Septum Perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal Septum Ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal Ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 4 | 3
Nausea (Gastrointestinal disorders) | 1 | 9 | 4 | 27 | 38
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 2
Nipple Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 4 | 3
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 5 | 5
Oesophageal Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Oral Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral Dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Oral Herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 4
Oral Mucosal Erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 8
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 6 | 13
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Otitis Externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis Media (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 6 | 14
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Palmar-plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 5 | 2 | 15 | 18
Palmoplantar Keratoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 3 | 2
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Periodontal Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Periorbital Oedema (Eye disorders) | 0 | 2 | 0 | 0 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 2
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Platelet Count Decreased (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 4
Prostatic Obstruction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0 | 15 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 4 | 1 | 4 | 10
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 6 | 12
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 6
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3
Red Blood Cells Urine (Investigations) | 0 | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Retinal Vein Occlusion (Eye disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 5
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Scrotal Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2
Sinus Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 6 | 3
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin Erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sternal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 3 | 8 | 18
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Swollen Tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 3
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 1 | 5
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5
Temperature Intolerance (General disorders) | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3
Thrombophlebitis Superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thyroid Disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Tinea Cruris (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tinea Pedis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Tinea Versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 3
Tooth Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 3
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 4 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 3 | 1
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 0 | 0 | 1 | 8 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Upper-airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Urethral Meatus Stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 2
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 3 | 4 | 5
Urinary Tract Pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Vaginal Lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 4 | 2
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 0 | 2
Vitamin D Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5 | 4 | 14 | 30
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulvovaginal Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Wandering Pacemaker (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 3 | 2 | 17 | 27
Weight Increased (Investigations) | 0 | 1 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
White Blood Cells Urine (Investigations) | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gait Disturbance (General disorders) | 1 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Speech Disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Duodenditis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Nasal Vestibulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pneumonial Staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Preventative Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Upper-airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Ear Haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of efficacy therefore protein biomarkers (P1b and P2), PK (P2), immunogenicity (P2) and disease control rate at 16 weeks by RECIST 1.1 and Choi criteria were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT01806064/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT01806064/SAP_001.pdf